CLINICAL TRIAL: NCT06980233
Title: Reentry-Assist App Development for Individuals With Addiction and Mental Illness
Brief Title: Reentry Assist (R-Assist)
Acronym: R-Assist
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meaningful Measurement, Inc (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001884; R41DA061403 (NIH)
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Substance Use Disorder (SUD); Mental Health Disorder; Criminal Recidivism
Keywords: substance use disorder; mental health; criminal-legal involvement
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders; Recidivism; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: R-Assist features will include: 1) daily self-reported symptom and medication management monitoring; 2) a 29-session MISSION-CJ self-help curriculum, with an accompanying library of recovery resources to support COD symptom management and promote prosocial thinking and behavior; 3) SDOH resource finder; and 4) a dashboard to track R-Assist engagement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-Assist (Experimental): Participants who have recently released from jail will engage with the R-assist app for up to 1.5 months
  Interventions: Behavioral: reentry assistance mobile health app

INTERVENTIONS:
Behavioral: reentry assistance mobile health app — R-Assist features will include: 1) daily self-reported symptom and medication management monitoring; 2) a 29-session MISSION-CJ self-help curriculum, with an accompanying library of recovery resources to support COD symptom management and promote prosocial thinking and behavior; 3) SDOH resource finder; and 4) a dashboard to track R-Assist engagement.

SUMMARY:
This project will aim to develop and pilot test, R-Assist, a mobile health application to support individuals with co-occurring substance use and mental health disorders (COD) in their recovery, who have recently released from a participating Massachusetts jail.

DETAILED DESCRIPTION:
This Phase I project will develop and test an mHealth app called R-Assist among individuals with COD recently released from a Massachusetts jail. R-Assist will offer four core features, including linkages to community resources via the resource locator, on demand, tailored self-help materials, and self-management/organizational tools. The following two Aims will be tested: Aim 1. R-Assist software and content prototype development. The 4 R-Assist features will include: 1) daily self-reported symptom and medication management monitoring; 2) a 29-session self-help curriculum, with an accompanying library of recovery resources to support COD symptom management and promote prosocial thinking and behavior; 3) social determinants of health (SDOH) resource finder; and 4) a dashboard to track R-Assist engagement. Aim 2. A successive cohort study of the R-Assist prototype with participants who have recently left jail (N = 38). This will include three successive field focus group cohorts with 18 participants, followed by a small open pilot with 20 participants. This project's four milestones will be executed in preparation for a larger Phase II trial.

* Milestone 1 (Months 1-5): R-Assist App Development and Interface Designs

  o No human subjects involvement
* Milestone 2 (Months 6-7): Initial Evaluation/Refinement of R-Assist

  o To recruit N=18 individuals for this Milestone
* Milestone 3 (Months 8-10): Open Pilot of R-Assist

  o To recruit recruit N=20 individuals for this Milestone
* Milestone 4 (Months 11-12): Product Refinement Prior to Phase II and Dissemination o No human subjects involvement

ELIGIBILITY:
Inclusion Criteria:

* Have been released from the participating jail within the past 150 days
* Own a smartphone (Android or iOS; 90% met this criterion in our prior studies)
* Have COD: any substance use disorder (we will allow poly-substance use disorders) and a co-occurring mental health disorder (depression, anxiety, trauma related disorders, bipolar, and/or schizophrenia)
* Consent to R-Assist app use observation and e-tracking
* Consent to audio recording during interviews and focus groups.

Exclusion Criteria:

* Acutely suicidal, homicidal, or psychotic
* Unable to provide informed consent
* Individuals released with monitoring devices or individuals involved in drug treatment courts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
App usage | From enrollment for 1.5 months during the open pilot
  Total time engaged in app will be tracked daily during open pilot period. Additionally, engagement and time with each feature will be tracked
System Usability Scale (SUS) | From enrollment for 1.5 months during the open pilot
  Overall score will be computed, indicating overall usability Score ranges from 0-100 (0-64=not acceptable, 65-84=acceptable, and 85, 100=excellent.
Mobile Application Rating Scale (MARS) | From enrollment for 1.5 months during the open pilot
  Overall score will be computed, indicating overall acceptability, as well as score for each of the four dimensions. The rating scale assesses app quality on four dimensions (1. Engagement, 2. Functionality, 3. Aesthetics, and 4. Information). All items are rated on 5-point scale from "1=inadequate" to "5=excellent"
Composite International Diagnostic Instrument for DSM-IV: Social determinants of health (SDOH) linkages | From enrollment for 1.5 months during the open pilot
  SDOH needs (e.g., housing instability, food insecurity, NA/AA/ other recovery linkages) will be assessed and the App will track all referrals and SDOH linkages made. Percent of linkages made to needed SDOH services will be examined.
Composite International Diagnostic Instrument for DSM-IV: Substance Use Disorder | From enrollment for 1.5 months during the open pilot
  Substance use disorder symptoms will be tracked daily during the open pilot period.
Composite International Diagnostic Instrument for DSM-IV: Mental Health | From enrollment for 1.5 months during the open pilot
  Mental health symptoms will be tracked daily during the open pilot period.

CONTACTS AND LOCATIONS:
Overall Officials: David Smelson, PsyD, Principal Investigator — University of Massachusetts Chan Medical School; Donna Surges Tatum, PhD, Principal Investigator — Meaningful Measurement, LLC

IPD SHARING:
Plan to Share IPD: No